CLINICAL TRIAL: NCT01900548
Title: Effect of Intake of Protein High in Ketogenic Amino Acids (e.g. Leucine) in Elderly Osteopenic Patients. Implications for Muscle, Bone , Metabolism, and Physical Function.
Brief Title: Effect of Intake of Whey Protein in Elderly Osteopenic Patients. Implications for Metabolism and Physical Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Council for Strategic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-136-13
Record Dates: First submitted 2013-06-10; First posted 2013-07-16 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2013-07

CONDITIONS: Osteopenia
Keywords: Osteopenia; Sarcopenia; Osteoporosis; Physical function; Body composition; Muscle protein; Leucine; Ketogenic amino acids; Resistance Training; Whey protein; Soy protein; Bone turnover
MeSH Terms: conditions — Bone Diseases, Metabolic; Sarcopenia; Osteoporosis | interventions — Whey Proteins; Soybean Proteins; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey protein (HPHL) (Experimental): Whey protein supplementation and resistance training for four month.
  Interventions: Dietary Supplement: Whey protein (HPHL); Other: Resistance training
- Soy protein (HPLL) (Experimental): Soy protein supplementation and resistance training for four month.
  Interventions: Dietary Supplement: Soy protein (HPLL); Other: Resistance training
- Placebo (P) (Placebo Comparator): Maltodextrin supplementation and resistance training for four month.
  Interventions: Dietary Supplement: Placebo (P); Other: Resistance training

INTERVENTIONS:
Dietary Supplement: Whey protein (HPHL) — The Whey protein group are supplemented 45 gram of whey protein, high protein high leucine (HPHL), every day.
  Arms: Whey protein (HPHL)
Dietary Supplement: Soy protein (HPLL) — The Soy protein group are supplemented 45 gram of Soy protein, high protein low leucine (HPLL), every day.
  Arms: Soy protein (HPLL)
Dietary Supplement: Placebo (P) — Will not be given protein but the same energy content using maltodextrin (in a blended fashion).
  Arms: Placebo (P)
Other: Resistance training — For 45 minutes 3 times a week the participants will complete resistance training with elastic bands in their own homes.

SUMMARY:
The aim of this study is to investigate potential metabolic effects of whey protein high in protein and high in leucine(HPHL) compared to soy protein high in protein and low in leucine(HPLL) in osteopenic patients in a randomized controlled intervention study.

The investigator hypothesize that HPHL will increase physical function and the ratio muscle mass / fat mass in this condition.

DETAILED DESCRIPTION:
With an increase in the older population in Denmark and most other countries there is an increase in the rate of patients with age related bone and muscle weakness. Proteins with a high content in ketogenic amino acids e.g. leucine have been investigated in relation to these conditions. Generally acute studies in animals and some in human have been conducted and have demonstrated positive effects in relation to prevention and treatment of bone and muscle weakness. We want to investigate these tendencies with supplementation of proteins in a randomized, blinded, 4 month intervention study with three arms - 1) the control group. 2) soy protein(high protein, low leucine). 3) Whey protein(high protein, high leucine). To increase any possible effect of the supplementation the subjects will complete a resistance training program concurrently. The study will focus on the anabolic properties of the ketogenic amino acids in animal whey protein compared to vegetable soy protein.

The investigator will study changes in:

* Gait speed related to muscle strength
* Walk distance in a Six-minute walk test related to sub maximal physical capacity
* Body composition (LBM/FM ratio) by a DEXA-scanner
* Biochemical markers on bone metabolism
* Bone-mineral-density(BMD) and -content(BMC)(DEXA scans)
* Muscle strength
* Body balance
* Protein and amino acid balance
* Nitrogen balance
* Gene-expression in muscle tissue
* Biochemical markers on fat- sugar- and protein-metabolism
* Biochemical markers on inflammation
* Blood pressure
* Insulin sensitivity by HOMA index
* Estimated maximal physical capacity by a bicycle ergometer test.

The perspective in this study is to develop a nutritional supplement with a high content of ketogenic amino acids (e.g. Leucine) that can be useful and beneficial in treatment and prevention of patients with bone and muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

* Osteopenia defined as BMD T-score <-1

Exclusion Criteria:

* Vitamin D deficiency defined as 25-hydroxyvitamin D (25-OH-D) below 30 nmol/l.
* Liver and kidney disease.
* Known diabetes or Hgb1c ≥6,5% (≥48mmol/l).
* Severe heart disease (NYHA-Class >2).
* Oral corticosteroid treatment within the last 3 month.
* Anamnestic information of hip fracture or vertebral fracture.
* Any antiosteoporotic treatment.
* participation in other intervention studies within the last 4 weeks.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
4 meter gait speed | Baseline and 4 months
  We will measure changes in 4 meter gait speed.
Walk distance | Baseline and 4 months
  We will measure changes in walk distance with the Six-Minute Walk Test.
Lean body mass(LBM)/Fat mass (FM) ratio. | Baseline and 4 months
  We will measure changes in the ratio LBM/FM with a DEXA-scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, Professor, Principal Investigator — The department of endocrinology, Aarhus University Hospital
Locations (1):
- Department of endocrinology, Aarhus University hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No